CLINICAL TRIAL: NCT02598882
Title: Physical Activity With an Active Video Game Provides Bigger Energy Expenditure and Less Muscle Fatigue
Brief Title: Virtual Reality as a Tool for Rehabilitation on Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daysi Tobelem, Principal investigator, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ExerRehab
Record Dates: First submitted 2015-10-16; First posted 2015-11-06 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Aged
Keywords: Elderly; Videogame; energy expenditure; electromyography; rehabilitation
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treadmill (Active Comparator): patients will be 30 minutes of activity on treadmill, before and after exercise the same shall be assessed as fatigue of quadriceps by surface electromyography
  Interventions: Device: treadmill
- videogame (Active Comparator): patients will be 30 minutes of activity with video games, before and after exercise the same shall be assessed as fatigue of quadriceps by surface electromyography
  Interventions: Device: videogame

INTERVENTIONS:
Device: videogame — Patients will be an assessment of quadriceps muscle strength by surface electromyography, before and after a 30-minute guided activity through an active video game
  Other Names: exergame; virtual reality
  Arms: videogame
Device: treadmill — Patients will be an assessment of quadriceps muscle strength by surface electromyography, before and after a 30-minute activity in treadmill.
  Arms: treadmill

SUMMARY:
Assessment of energy expenditure and the quadriceps muscle fatigue of healthy seniors, after two physical activities, being one of an activity guided by interactive video game (Xbox) and another on the treadmill. The participants will perform the activities in two different days, the order will be obtained by randomization.

ELIGIBILITY:
Inclusion Criteria:

* Participate in this study elderly
* Of both sexes,
* Over 60 years,
* without cardiac and respiratory diseases
* Who accept to participate in the research, giving your consent by signing the informed consent

Exclusion Criteria:

* Those who oppose the signing of the informed consent
* Submit proposals and activities intolerance who can't understand or accomplish correctly the procedures due to physical and or mental limitations.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Assessment of quadriceps muscle fatigue | one year

SECONDARY OUTCOMES:
Evaluation of heart rate's | one year
  during the activities the patients will be evaluated as the heart rate variation, by means of a frequency meter
Evaluation of peripheral oxygen saturation | one year
  During the activities the patients will be evaluated as the peripheral oxygen saturation, by means of a Pulse Oximeter.
Assessment of energy expenditure | one year
  during the implementation of the proposed activities, patients will be assessed to the energy expenditure with the use of an armband

CONTACTS AND LOCATIONS:
Overall Officials: Dirceu Costa, Doctor, Study Director — University of Nove de Julho
Locations (1):
- Dirceu Costa, São Paulo, Brazil